CLINICAL TRIAL: NCT01552733
Title: Robotic Therapy Early After Stroke Events
Acronym: R-TEASE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NHS Greater Glasgow and Clyde (Other)
Collaborators: University of Glasgow (Other)
Responsible Party: Principal Investigator, Dr Jesse Dawson, Clinical Senior Lecturer in Medicine / Honorary Consultant, University of Glasgow
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GN12MT023; R12/A141 (Other Grant/Funding Number: Chest Heart and Stroke Scotland)
Record Dates: First submitted 2012-03-09; First posted 2012-03-13 (Estimated); Last update posted 2017-01-27 (Estimated); Status verified 2017-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke | interventions — Standard of Care

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Robotic Therapy (Experimental): Robotic Therapy using 'Inmotion' device plus standard care. Participants randomised to robotic therapy will receive up to 12 sessions (approximately 1 hour each) performing tasks (including circle drawing, reaching targets and holding/moving against moderate resistance.
  Interventions: Device: 'Inmotion Arm Robot'
- Standard Care (Placebo Comparator): Rehabilitation therapy according to local guidelines.
  Interventions: Other: Standard of care

INTERVENTIONS:
Device: 'Inmotion Arm Robot' — To improve limb function in those with limb impairment
  Arms: Robotic Therapy
Other: Standard of care — Rehabilitation Therapy
  Arms: Standard Care

SUMMARY:
Weakness and impairment of the upper limb is a common contributing factor to post stroke disability. Specially designed robotic systems have been developed to try to improve this. The investigators already know that their use helps improve limb function after stroke when it has been present for many months. The investigators do not know whether they can help early after stroke and enhance recovery of limb function, and perhaps prevent weakness becoming chronic.

The investigators plan a randomised controlled blinded study to explore the benefits of robot assisted therapy early after stroke in 80 stroke survivors. Participants will be randomised by 7 days after stroke to standard care or to robotic therapy (40 participants per study group).

Standard of care will be rehabilitation therapy according to local guidelines delivered by NHS multidisciplinary team.

Robotic therapy sessions lasts approximately one hour and consists of a series of tasks in first the unimpaired then impaired limb. The robotic-assisted therapy will consist of a series of taks including circle-drawing, reaching targets and holding/moving against moderate resistance. Twelve sessions of therapy within the first 4 weeks after randomisation will be delivered. This study will take 3 years to complete.

ELIGIBILITY:
Inclusion Criteria:

1. Aged > 18 years
2. Confirmed diagnosis of stroke
3. Randomisation by seven days
4. Upper limb impairment, defined as a measurable upper limb impairment on the NIHSS and a baseline upper limb FuglMeyer score of <50 at randomisation
5. Able to comply with the requirements of the protocol

Exclusion Criteria:

1. Other significant upper limb impairment e.g. fixed contracture, fracture, frozen shoulder, severe arthritis, amputation.
2. Diagnosis likely to interfere with rehabilitation or outcome assessments such as registered blind or terminal illness.
3. Participation in other stroke rehabilitation trial.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2012-03-01 (Actual); Primary Completion 2016-03-16 (Actual); Study Completion 2016-03-16 (Actual)

PRIMARY OUTCOMES:
Fugl-Meyer score therapy. | One month
Feasibility | One month
  Defined as the proportion of individuals randomised to robotic intervention who complete 12 sessions of Robotic therapy. Will serve as a coprimary endpoint.

SECONDARY OUTCOMES:
Fugl-Meyer score. | Day 90
Modified Rankin scale score | DAy 90
Barthel index | Day 90
Stroke Impact Scale | Day 90
NIHSS | Day 90
Action Research Arm Test | Day 90

CONTACTS AND LOCATIONS:
Overall Officials: Jesse Dawson, MD, Principal Investigator — University of Glasgow
Locations (1):
- Western Infirmary, NHS Greater Glasgow and Clyde, Glasgow, United Kingdom